CLINICAL TRIAL: NCT06552364
Title: Air Pollution and Inhaled Corticosteroids in COPD
Acronym: APIC
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: University of Calgary (Other); University of Ottawa (Other); University of Manitoba (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Christopher Carlsten, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: H22-03008
Record Dates: First submitted 2024-03-28; First posted 2024-08-14 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: COPD
Keywords: Air Pollution; Inhaled Corticosteroid; LABA/LAMA; Triple Therapy (LABA/LAMA/ICS)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Vehicle Emissions

STUDY DESIGN:
Intervention Model Description: Participants will become their own control as they experience all four combinations of exposures at four different time intervals, each separated by at least a month for washout: 1) Filtered Air-Inhaled Corticosteroid (FA-ICS), 2) Filtered Air- No Inhaled Corticosteroid (FA-no ICS), 3) Diesel Exhaust-Inhaled Corticosteroid (DE-ICS), and 4) Diesel Exhaust- No Inhaled Corticosteroid (DE-no ICS).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding of exposures will be performed by the air pollution exposure laboratory (APEL) engineer. Visually indistinguishable inhalers will be coded by research pharmacy staff. All assays will be performed by personnel who do not know the exposure conditions of individual samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Filtered Air with LABA/LAMA (Placebo Comparator): Participants will inhale a ultra Long-Acting Beta-Agonist (LABA; vilanterol (25mcg)) + Long-acting Muscarinic Antagonist (LAMA; umeclidinium (62.5mcg)) combination medication once daily for 28+ days before sitting in a booth and being exposed to high-efficiency particulate air (HEPA) filtered air for 2 hours.
  Interventions: Drug: LABA+LAMA; Other: Filtered Air
- Filtered Air with LABA/LAMA + ICS (Active Comparator): Participants will inhale a LABA (vilanterol (25mcg)) + LAMA (umeclidinium (62.5mcg))+ Inhaled Corticosteroid (ICS; fluticasone furoate (100mcg)) medication once daily for 28+ days before sitting in a booth and being exposed to HEPA-filtered air for 2 hours.
  Interventions: Drug: LABA+LAMA+ICS; Other: Filtered Air
- Diesel Exhaust with LABA/LAMA (Active Comparator): Participants will inhale a LABA (vilanterol (25mcg)) + LAMA (umeclidinium (62.5mcg)) medication once daily for 28+ days before sitting in a booth and being exposed to diesel exhaust (standardized to 300µg/m³ of particulate matter with a diameter of 2.5 micrometers or less (PM2.5)) for 2 hours.
  Interventions: Drug: LABA+LAMA; Other: Diesel Exhaust
- Diesel Exhaust with LABA/LAMA + ICS (Experimental): Participants will inhale a LABA (vilanterol (25mcg)) + LAMA (umeclidinium (62.5mcg))+ Inhaled Corticosteroid (ICS; fluticasone furoate (100mcg)) medication once daily for 28+ days before sitting in a booth and being exposed to diesel exhaust (300ug/m3 of PM2.5) for 2 hours.
  Interventions: Drug: LABA+LAMA+ICS; Other: Diesel Exhaust

INTERVENTIONS:
Drug: LABA+LAMA — 1 dose per day (AM)
  Other Names: Anoro Ellipta
  Arms: Diesel Exhaust with LABA/LAMA; Filtered Air with LABA/LAMA
Drug: LABA+LAMA+ICS — 1 dose per day (AM)
  Other Names: Trelegy Ellipta
  Arms: Diesel Exhaust with LABA/LAMA + ICS; Filtered Air with LABA/LAMA + ICS
Other: Filtered Air — Exposure to HEPA filtered air, as a control
  Arms: Filtered Air with LABA/LAMA; Filtered Air with LABA/LAMA + ICS
Other: Diesel Exhaust — Diesel exhaust standardized to 300µg/m³ of particulate matter with a diameter of 2.5 micrometers or less (PM2.5).
  Other Names: Traffic Related Air Pollution
  Arms: Diesel Exhaust with LABA/LAMA; Diesel Exhaust with LABA/LAMA + ICS

SUMMARY:
Studies have shown that people with chronic obstructive pulmonary disease (COPD) have worse symptoms after breathing polluted air. People with COPD also often need to go to the hospital if they get a virus or other bug. One of the main drugs taken for COPD treatment (inhaled corticosteroid) may change COPD patients' lungs in ways that make it harder to deal with bugs, especially if they breathe in polluted air. If so, this could cause more frequent hospital visits. On the other hand, the same drug (inhaled corticosteroid) helps some people control symptoms, and may help them avoid hospital visits. The APEL investigators are conducting this study (APIC) to understand if this drug (inhaled corticosteroid), in combination with polluted air, will change the lungs of those with COPD in ways that make it more likely to catch bugs or have other problems.

DETAILED DESCRIPTION:
APIC will involve 48 volunteer participants (24 of each biological sex assigned at birth) with mild-to-moderate COPD where the researchers will look at what (if any) are the differences between breathing in fresh air (filtered air - FA) or polluted air (diesel exhaust - DE) while taking the drug (Inhaled corticosteroid - ICS) or not (no ICS), both in combination with two standard COPD medicines that make it easier to breath (a long-acting beta-agonist and a long-acting muscarinic antagonist). The participant will take an inhaled medication daily throughout the study. This study will use a controlled amount of diesel exhaust to model traffic-related air pollution (TRAP), a commonly encountered form of polluted air.

Each participant will act as their own control, as they will experience all four combinations: 1) FA-ICS, 2) FA-no ICS, 3) DE-ICS, and 4) DE-no ICS. These combinations will be randomized in what researchers call a double-blinded crossover study, so that every participant will get these combinations in a different order. However, only the engineer on the team will be allowed to know which participant gets what. Blinding will prevent everyone else, including the participant, from being biased against the conditions and affecting outcomes based on this perception.

The study will span over five months (approximately 121 days of active commitment), which includes ten in-person visits to a research office at the Vancouver General Hospital, for a total of approximately 40 hours. While the participant is on-site, the investigators will supervise a series of questionnaires, sample collection (blood, urine, bronchoscopy lung samples), and lung function tests. The investigators will evaluate multiple endpoints as detailed in the Outcome Measures section. For each applicable endpoint, the investigators will evaluate stratified analyses and effect modification by biological sex, participant age, gene score, and microbiomes.

The investigators do not expect that the participant's responses to either the corticosteroid or diesel exhaust will be noticeable to them. Any responses that may occur will probably only be detectable through careful examination of their cells and tissues (e.g., blood, urine, bronchial samples). However, understanding the subtle changes that may occur could help reduce or prevent health problems associated with TRAP exposure in the future.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 40 to 80
* Mild-to-moderate COPD diagnosis (Global Initiative for Chronic Obstructive Lung Disease stage 1-2) as confirmed by medical history, questionnaires, and spirometry (a test that measures the amount of air one can breathe in and out of the lungs) results
* Spirometry results will be assessed by the study physician to determine eligibility

Exclusion Criteria:

* Currently smoking or have been smoking within six months of your screening visit for this study
* Have had an acute exacerbation of COPD (AECOPD) diagnosis within 365 days of the screening visit
* Have a history of asthma or asthma-COPD overlap syndrome
* Existing medical condition or other health concerns as assessed by the study physician
* Pregnant, plan to be pregnant, or breastfeeding during your enrolment in the study. Participants of childbearing potential will be required to have a negative pregnancy test prior to study inclusion.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Inhaled corticosteroid (ICS) and/or diesel exhaust exposure effects on inflammatory cells. | Comparison of the different arms over the span of 5 months.
  Differentially count lung cells.
Inhaled corticosteroid (ICS) and/or diesel exhaust exposure effects on exhaled nitric oxide. | Comparison of the different arms over the span of 5 months.
  Measurement of fractional exhaled nitric oxide (FeNO).
Inhaled corticosteroid (ICS) and/or diesel exhaust exposure effects on anti-microbial host defense proteins. | Comparison of the different arms over the span of 5 months.
  Anti-microbial host defense (AMP) matrix, determined from, for example, human neutrophil peptide 1 (HNP1; DEFA1), calprotectin (S100A8/S100A9), cathelicidin antimicrobial peptide/LL-37, Lipocalin-2 (LCN2), and S100 calcium-binding protein A7 (S100A7) in the lungs. And dermcidin (DCD), calprotectin (S100A8/S100A9), cathelicidin antimicrobial peptide/LL-37, and amphiregulin (AREG) in peripheral blood.
Inhaled corticosteroid (ICS) and/or diesel exhaust exposure effects on oxidative stress in the lungs. | Comparison of the different arms over the span of 5 months.
  Determine oxidative stress (e.g. H2DCFDA) in the lungs.
Inhaled corticosteroid (ICS) and/or diesel exhaust exposure effects on neutrophil extracellular TRAPs (NETs). | Comparison of the different arms over the span of 5 months.
  Analysis of counts of neutrophil extracellular TRAPs (NETs).
Inhaled corticosteroid (ICS) and/or diesel exhaust exposure effects on lung inflammatory markers. | Comparison of the different arms over the span of 5 months.
  An inflammation matrix will be generated, including data from RNA and proteins (e.g. serum amyloid A (SAA), c-reactive protein (CRP), chemokine ligand 18 (CCL18) and fibrinogen), in the lungs.

SECONDARY OUTCOMES:
Inhaled corticosteroids (ICS) and/or diesel exhaust exposure induced modulation of circulating markers of inflammation. | Comparison of the different arms over the span of 5 months.
  An inflammation matrix will be generated, including data from RNA and proteins (e.g., CRP, CCL18, fibrinogen, CX3CL1, CCL23, CXCL8, SAA, MMP9, MMP12, APOB, APOM) in peripheral blood.
Inhaled corticosteroid (ICS) and/or diesel exhaust exposure induced modulation of circulating cells and inflammatory cellular markers. | Comparison of the different arms over the span of 5 months.
  Measurement of cellular inflammation scores from complete cell counts, and cellular markers (e.g. CD80, CD86, HLA-DR, CD283, CD288, CD119, TLR7, CD16, CD64, CD11b, CD206, CXCR2) in peripheral blood.
Inhaled corticosteroid (ICS) and/or diesel exhaust exposure induced modulation of lung resistance as assessed by oscillometry. | Comparison of the different arms over the span of 5 months.
  Lung resistance and reactivity from respiratory oscillometry Rrs5, Rrs20, Rrs5-20, Xrs5, AX and Fres.
Inhaled corticosteroid (ICS) and/or diesel exhaust exposure effects on lung function. | Comparison of the different arms over the span of 5 months.
  Lung function as evaluated by spirometry (e.g. FEV1).
Effects of inhaled corticosteroids (ICS) and/or diesel exhaust on neutrophil function. | Comparison of the different arms over the span of 5 months.
  Neutrophil respiratory burst (Fc-OxyBURST Green) measurement.
Effects of inhaled corticosteroids (ICS) and/or diesel exhaust on phagocytosis. | Comparison of the different arms over the span of 5 months.
  Measurement of phagocytosis (fluorescein isothiocyanate-labelled opsonized S. cerevisiae zymosan-A bioparticles uptake).
Effects of inhaled corticosteroids (ICS) and/or diesel exhaust on the EXACT (and E-RS:COPD) questionnaire. | Comparison of the different arms over the span of 5 months.
  The EXACT (and its derivative instrument E-RS (Evaluating Respiratory Symptoms):COPD) questionnaire (see https://www.evidera.com/what-we-do/patient-centered-research/coa-instrument-management-services/exact-program/exact-content/) will be completed.
Effects of inhaled corticosteroids (ICS) and/or diesel exhaust on the mMRC dyspnea scale questionnaire. | Comparison of the different arms over the span of 5 months.
  The modified Medical Research Council (mMRC) Dyspnea Scale (see https://www.pcrs-uk.org/mrc-dyspnoea-scale) will be completed.
Effects of inhaled corticosteroids (ICS) and/or diesel exhaust on the Symptoms and Perception questionnaire. | Comparison of the different arms over the span of 5 months.
  The Symptoms and Perception questionnaire (see https://particleandfibretoxicology.biomedcentral.com/articles/10.1186/s12989-022-00506-6#Sec15) will be completed.
Effects of inhaled corticosteroids (ICS) and/or diesel exhaust on the Perceived Stress Scale questionnaire. | Comparison of the different arms over the span of 5 months.
  The Perceived Stress Scale questionnaire (see https://www.das.nh.gov/wellness/docs/percieved%20stress%20scale.pdf) will be completed.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Carlsten, MD, MPH, Principal Investigator — University of British Columbia; Neeloffer Mookherjee, PhD, Principal Investigator — University of Manitoba; Shawn Aaron, MD, FRCPC, Principal Investigator — University of Ottawa/Université d'Ottawa; Janice Leung, MD, FRCPC, Principal Investigator — University of British Columbia; Christopher F Rider, PhD, Principal Investigator — University of British Columbia; Neil Alexis, PhD, Principal Investigator — University of North Carolina, Chapel Hill